CLINICAL TRIAL: NCT04668911
Title: Oral Health, Microbial Burden and COVID-19
Acronym: ORACLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eastman Dental Insitute and Hospital (Other)
Collaborators: DermBiont, Inc. (Industry); University College London Hospitals (Other); The Whittington Hospital NHS Trust (Other Government)
Responsible Party: Principal Investigator, Prof Francesco D'Aiuto, Professor, University College, London
Other Study IDs: EDGE 132868; 283766 (Other: IRAS)
Record Dates: First submitted 2020-12-11; First posted 2020-12-16 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Periodontitis
Keywords: COVID-19; Human microbiome; Oral microbiome; SARS-CoV-2 infection
MeSH Terms: conditions — COVID-19; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Oral and nasal swab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Controls tested PCR (-) for COVID-19
  Interventions: Other: Swab
- Tested PCR (+) for COVID-19, Mild - not admitted to the hospital
  Interventions: Other: Swab
- Tested PCR (+) for COVID-19, Severe - admitted to ICU (Intensive Care Unit)
  Interventions: Other: Swab

INTERVENTIONS:
Other: Swab — PCR test for SARS-CoV2, oral and nasal swab

SUMMARY:
An observational study of patients with COVID-19 confirmed cases (with various degrees of severity) and controls.

Oral and nasal swabs will be taken from 150 patients (50 with mild form and 50 with severe form of COVID-19 with or without mechanical ventilation, 50 healthy controls).

ELIGIBILITY:
Inclusion Criteria:

1. Must provide written informed consent
2. Subjects have to be tested (PCR) positive or negative for SARS-CoV2 infection
3. Must be able to provide oral and nasal swabbing within 48 hours of polymerise chain reaction (PCR) test results

Exclusion Criteria:

a. Under the age of 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults who tested (PCR) positive or negative for SARS-CoV2 infection
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-12-13 (Actual); Primary Completion 2021-12-12 (Estimated); Study Completion 2021-12-12 (Estimated)

PRIMARY OUTCOMES:
Oral microbial signature | Day 1
  To assess the oral microbial signatures that relates to SARS-CoV2 in patients with no, mild and severe disease.

SECONDARY OUTCOMES:
Nasal microbial signature | Day 1
  To assess the nasal microbial signatures related to SARS-CoV2 in patients with no, mild and severe disease and to assess the role of the oral expression of ACE2-Ang II system during SARS-CoV2 in relation to disease outcome (mild, severe COVID).

CONTACTS AND LOCATIONS:
Locations (1):
- University College Hospital (UCH), UCL Eastman Dental Institute, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided